CLINICAL TRIAL: NCT06014164
Title: Qualitative Study of the Self-administered Therapeutic Use of Psychedelics in People With Psychiatric Disorders
Brief Title: Qualitative Study About Psychedelics Using in Psychiatric Disorders
Acronym: PSYCHEQUALI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0396; 2023-A01575-40 (Other: ID-RCB)
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Psychiatric Disorder
Keywords: Psychiatric disorder; Psychedelics
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients using psychedelic substances: Adult patients self-administering psychedelic substances in psychiatric disorders
  Interventions: Diagnostic Test: Interview

INTERVENTIONS:
Diagnostic Test: Interview — An interview will be conducted to describe the experiences of people with psychiatric disorders who use psychedelic substances for therapeutic purposes

SUMMARY:
This study is set up to better understand the current use of psychedelics in France in the general population. The present focus on individuals who have used any type of psychedelic drug in order to suppress or alleviate a psychiatric symptom in the context of a diagnosed pathology. The data are collected during a semi-structured interview and then studied in a thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a psychiatric disorder by a psychiatrist or general practitioner
* Patients used psychedelic or related substances in order to treat psychiatric symptoms
* Patients have given their oral non-opposition
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Patients who don't speak or understand French
* Patients under protection, guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients self-administering psychodelic substances for therapeutic purposes
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Experiences of people using psychedelic substances | Baseline
  Experiences description of people with psychiatric disorders who use psychedelic substances for therapeutic purposes will be assessed by interview

SECONDARY OUTCOMES:
Profile of people using psychedelic substances | Baseline
  The profile of people with psychiatric disorders who use psychedelic substances for therapeutic purposes will be assessed by interview

CONTACTS AND LOCATIONS:
Overall Officials: Antoine YRONDI, MD, Principal Investigator — University Hospital, Toulouse